CLINICAL TRIAL: NCT02503579
Title: What's the Role of Brain-derived Neurotrophic Factor in the Relationship Between Executive Function and Physical Fitness/Training in Typically Developing Children? A Randomized Controlled Study
Brief Title: The Role of Brain-derived Neurotropic Factor in the Relationship Between Executive Function and Physical Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2015/0520
Record Dates: First submitted 2015-05-29; First posted 2015-07-21 (Estimated); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Executive Dysfunction; Motor Activity; Child
Keywords: Brain-derived neurotropic factor; Executive function
MeSH Terms: conditions — Motor Activity | interventions — Physical Conditioning, Human

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- physical training (Experimental): Participant receive a submaximal (60% -75% maximal oxygen uptake) physical activity training of 30 minutes during 8 weeks, 2 times a week. Individual heart rates will be monitored during the training.
  Interventions: Behavioral: physical training
- control (No Intervention): 1 training at the beginning of the study
  1 training at the end of the study

INTERVENTIONS:
Behavioral: physical training — physical activity program, 30 minutes
  Arms: physical training

SUMMARY:
This doctoral thesis has the aim to identify the role of Brain-derived neurotropic factor in the relationship between physical fitness/activity and executive functions in typically developing children and children with Autism Spectrum Disorder, Development Coordination Disorder , Attention Hyperactive Disorder.

DETAILED DESCRIPTION:
Nowadays children are getting more inactive and participate less in sports or daily physical activity. Previous studies have shown that a good physical fitness is associated with improved cognitive functions. While being physical active, physiological changes take places in the brain. Brain-derived neurotropic factor is one of the neurotropins that plays a crucial role in this process. Executive functions are cognitive processes that are responsible for organizing and controlling goal-directed actions. These functions are developing during childhood and play an important role in daily- and school functioning.

This doctoral thesis has the aim to identify the role of Brain-derived neurotropic factor in the relationship between physical fitness/activity and executive functions in children.

In a first trail the effect of physical fitness and physical training on executive functioning and levels of Brain-derived neurotropic factor will be studied.

In a second trail the research question is expanded by investigating the same relations in children with Autism Spectrum Disorder, Development Coordination Disorder , Attention Hyperactive Disorder.

Protocol trail 1: The included (typically developing) children will be randomized and stratified for level of physical fitness into 2 groups: the intervention group and the control group. The intervention group will receive physical activity training 2 times a week during 8 weeks. The control group will receive no additional training. At the beginning and the end of the training period both the intervention and control group will be tested for physical fitness and level of executive functioning.

Protocol trail 2: Identical protocol to trail 1 except the participants will be children with Autism Spectrum Disorder, Development Coordination Disorder , Attention Hyperactive Disorder in stead of typically developing children.

ELIGIBILITY:
Trail 1

Inclusion Criteria:

* typically developing children

Exclusion Criteria:

* children with: executive function-, neurological- or cognitive disorders

Trail 2

Inclusion criteria:

* typically developing children (control)
* children with Developmental Coordination disorder, Attention deficit disorder or Autism Spectrum disorder

Exclusion criteria:

* Children with neurological- or cognitive disorders

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2015-08; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline after 9 weeks in concentration of serum brain-derived neurotropic factor in blood sample. | Baseline and change from baseline 9 weeks later.
  Measurement of serum Brain-derived neurotropic factor true blood samples.
Change from Baseline after acute physical activity in concentration of serum brain-derived neurotropic factor in blood sample | Baseline and change from baseline after 30 minutes of training.
  Measurement of serum Brain-derived neurotropic factor true blood samples.

SECONDARY OUTCOMES:
Change of baseline after 9 weeks in Amount of daily physical activity (hours/week) | Baseline and change from baseline 9 weeks later.
  Questionnaire about daily physical activity.
Change of baseline after 9 weeks in Maximal Oxygen Uptake during exertion test. | Baseline and change of baseline 9 week later.
  Physical fitness measurement with maximal endurance test on bicycle using Balke-protocol.
Change of baseline after 9 weeks in Maximal heart rate during exertion test. | Baseline and change of baseline 9 week later.
  Physical fitness measurement with maximal endurance test on bicycle using Balke-protocol.
Change from Baseline after 9 weeks on Executive functioning test battery. | Baseline and change of baseline 9 weeks later.
  EF measurement true computer tasks.
Change from Baseline after acute physical activity on Executive functioning test battery. | Baseline and change of baseline after 30 minutes of physical activity.
  EF measurement true computer tasks.

CONTACTS AND LOCATIONS:
Overall Officials: Hilde Van Waelvelde, Professor, Principal Investigator — Revaki

REFERENCES:
- [Derived] Latomme J, Calders P, Van Waelvelde H, Marien T, De Craemer M. The Role of Brain-Derived Neurotrophic Factor (BDNF) in the Relation between Physical Activity and Executive Functioning in Children. Children (Basel). 2022 Apr 22;9(5):596. doi: 10.3390/children9050596. PMID 35626772